CLINICAL TRIAL: NCT01710631
Title: A Randomized, Double-Blind, Placebo-Controlled and Open-Label Twelve Month Study of the Safety of (S)-Zopiclone in Adult Subjects With Insomnia
Brief Title: Twelve Month Study of the Safety of Eszopiclone in Adult Subjects With Insomnia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 190-049
Record Dates: First submitted 2012-10-17; First posted 2012-10-19 (Estimated); Last update posted 2012-10-22 (Estimated); Status verified 2012-10

CONDITIONS: Primary Insomnia
Keywords: Sleep
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Eszopiclone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- eszopiclone 3 mg (Experimental): eszopiclone 3 mg (comprised of either two 1.5 mg tablets, or one 1 mg tablet and one 2 mg tablet).
  Interventions: Drug: eszopiclone 3 mg
- placebo (Placebo Comparator): placebo tablet
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: eszopiclone 3 mg — eszopiclone 3 mg (comprised of either two 1.5 mg tablets, or one 1 mg tablet and one 2 mg tablet).
  Other Names: lunesta
  Arms: eszopiclone 3 mg
Drug: placebo — placebo
  Arms: placebo

SUMMARY:
A six-month study to determine the safety and efficacy with an additional open-label extension to determine the long-term safety of eszopiclone in the treatment of adult subjects with primary insomnia.

DETAILED DESCRIPTION:
A six month, randomized, double-blind and six month open-label extension, multi-center, outpatient study to determine the safety of eszopiclone in the treatment of adult subjects with primary insomnia. Approximately 800 subjects were to be randomized using a 3:1 ratio to receive one of the two treatments, eszopiclone 3 mg or placebo, for 6 months. All subjects completing 6 months of treatment were eligible to receive open-label 3 mg eszopiclone for an additional 6 months. Subjects were allowed to stay on study for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Subject met Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) criteria for primary insomnia and reported sleeping no more than 6.5 hours per night and/or taking more than 30 minutes each night to fall asleep for at least one month prior to screening.
* Subject was between 21 and 64 years of age (inclusive) at screening. Both males and females were eligible to participate.
* Subject provided written informed consent indicating that the purpose of the study was understood. The subject was willing to adhere to the regimen and study procedures described in this protocol.
* Females of childbearing potential must have willingly signed "Women of Child-Bearing Potential Informed Consent" addendum. Females considered not of childbearing potential must have been surgically sterile or greater than one-year post-menopausal, defined as a complete cessation of menstruation for at least one year.
* Subject's physical examination, including a brief neurological examination, showed no clinically significant abnormal findings at screening.
* Subject had no known clinically significant abnormal laboratory findings at screening.
* Subject had no clinically significant Electrocardiography (ECG) abnormalities at screening.

Exclusion Criteria:

* Subject had any clinically significant unstable medical abnormality, chronic disease, or a history of a clinically significant abnormality of the cardiovascular, respiratory, hepatic, or renal systems.
* Subject had a history of, or current malignancy except for non-melanomatous skin cancer.
* Subject had objective evidence of active thyroid disease at screening. Subjects on thyroid replacement therapy were included as long as dose had been stable for ≥ 3 months.
* Subject had a DSM-IV Axis I psychiatric diagnosis other than Sexual and Gender Identity Disorders, or Axis II Personality Disorders (but not schizotypal, schizoid, or borderline personality disorder). Other non-psychotic Axis I disorders except dementia and delirium were considered on a case-by-case basis.
* Subject had a known sensitivity to racemic zopiclone, any benzodiazepine, any sedative hypnotic, any substance that was contained in the formulation, or had been hospitalized for any allergic conditions (e.g. recurrent dermatitis, drug hypersensitivity, drug allergy, etc.).
* Subject had difficulties in sleep initiation or maintenance associated with known sleep difficulties (e.g. sleep apnea, restless leg syndrome, (RLS) or periodic leg movement syndrome (PLMS)), or had any condition which had, or may, affect sleep (e.g., chronic pain, Benign prostatic hyperplasia (BPH), etc.).
* Subject had history of substance abuse in the past 10 years or substance dependence at any time; positive urine drug test at screening.
* Subject tested positive at screening for hepatitis B surface antigen, hepatitis C antibody or had a history of a positive result.
* Subject was known to be seropositive for Human immunodeficiency virus (HIV).
* Female subjects who were pregnant, lactating or within 6 months post-partum.
* Subject had a disorder or history of a condition (e.g., malabsorption, gastrointestinal surgery) that may have interfered with drug absorption, distribution, metabolism, or excretion.
* Subject had used any drugs known or suspected to affect hepatic or renal clearance capacity within a period of 30 days prior to screening.
* Subject self-reported consumption of more than two alcoholic beverages daily, 14 or more alcoholic beverages weekly, or five or more alcoholic beverages on any given day.
* Subject had taken any psychotropic medications or other medications known to affect sleep within the 3 days prior to screening visit or was anticipated to need any of these types of medications during double-blind treatment.
* Subject had participated in any investigational study within 30 days prior to screening.
* Subject had taken herbal supplements, purported to have central nervous system effects, (tablets, powders, extracts or tinctures) or combination products with herbs or melatonin within 14 days prior to screening or St. John's Wort within 30 days prior to screening.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 791 (Actual)
Dates: Start 2001-02; Primary Completion 2002-08 (Actual); Study Completion 2002-08 (Actual)

PRIMARY OUTCOMES:
Average sleep latency over the last half of the double-blind study period ("last-three-month average" = mean of the monthly averages for months 4, 5, and 6) | Months 4-6
Occurrence of Adverse Events (AEs) to evaluate the safety of eszopiclone | 12 Months

SECONDARY OUTCOMES:
Subjective Total sleep time | Months 4-6 average
Subjective Sleep latency | Months 1-3
Number of awakenings | Months 1-12
Wake Time After Sleep Onset (WASO) | Months 1-12
Quality of Sleep | Months 1-12
AE's | 12 months
Total sleep time | Months 1-3

CONTACTS AND LOCATIONS:
Overall Officials: Lunesta Medical Director, MD, Study Director — Sumitomo Pharma America, Inc.